CLINICAL TRIAL: NCT05505383
Title: The Effect of Backward Walking Training on Balance, Gait and Functional Mobility in Patients With Multiple Sclerosis Patients
Brief Title: The Effect of Backward Walking Training on Balance, Gait and Functional Mobility in Patients With Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Saglik Bilimleri Universitesi (Other)
Collaborators: Ankara University (Other)
Responsible Party: Principal Investigator, Fatih Söke, Assistant Professor, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022/412
Record Dates: First submitted 2022-08-16; First posted 2022-08-17 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; backward walking training; balance; gait; functional mobility
MeSH Terms: conditions — Multiple Sclerosis | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Backward walking training group (Experimental): This group will participate in a backward walking training program (8-week, 3 times weekly, and 30-min each time) and conventional gait training program (8-week, 3 times weekly, and 45-min each time).
  Interventions: Other: Exercise training
- Conventional gait training (Active Comparator): This group will participate in a conventional gait training program (8-week, 3 times weekly, and 45-min each time).
  Interventions: Other: Exercise training

INTERVENTIONS:
Other: Exercise training — People with multiple sclerosis will be received a supervised physiotherapy and rehabilitation program.

SUMMARY:
Backward walking training can be a useful treatment approach, providing novel balance and gait challenges. It can lead to improve balance, gait and functional mobility in neurologic populations. However, the effect of backward walking training has net been investigated in people with multiple sclerosis.

DETAILED DESCRIPTION:
Multiple sclerosis is a chronic autoimmune disease of the central nervous system. Patients with multiple sclerosis have problems in balance, gait, and functional mobility. This problems can lead to falls, injuries, hospitalization, limited daily living activities, and decreased quality of life. Backward walking is a popular training approach to improve balance, gait, and functional mobility in other neurological disease such as stroke, and Parkinson's disease. Moreover, backward walking performance decreases in multiple sclerosis. However, no study has been performed to determine the effectiveness of backward walking training in multiple sclerosis. Therefore, this study aimed to investigate the effect of backward walking training on balance, gait, and functional mobility in patients with multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years,
* neurologist-diagnosed Multiple Sclerosis,
* Expanded Disability Status Scale (EDSS) score between 0 and 5.5,
* no MS exacerbation within the last 3 months,
* use of stable medication in the last 3 months,
* not received immunomodulator treatment within the last 6 months,

Exclusion Criteria:

* other neurologic disorder,
* Pregnancy,
* Cardiovascular, orthopedic, or systemic any disease hindering the participation of exercise program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2022-08-18 (Actual); Primary Completion 2022-11-20 (Estimated); Study Completion 2022-12-20 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Scale [Time Frame: 10 minutes] | 10 minutes
  Functional balance is assessed by using the Berg Balance Scale. During the test, participants are asked to perform 14 tasks frequently used in daily life activities. Each item is scored between 0 (unable to perform the task) and 4 (task is performed independently) according to the ability of the person while performing the task. The highest possible score is 56 points. A higher score indicates better balance.
Four Square Step Test | 15 seconds
  The Four Square Step Test measures dynamic balance and clinically assesses the person's ability to step over objects forward, sideways, and backward. A square was formed by 4 canes resting flat on the floor. The participants were instructed to try and complete the sequence as fast as possible without touching the canes with both feet, making contact with the floor in each square.
Activities-specific Balance Confidence Scale | 2 minutes
  Participants are asked to rate their balance confidence level 0% and 100% in the 16-item related to various everyday activities. The mean score on the 16-item questionnaire ranges from 0 to 100% and higher scores indicate a better balance confidence.
10 Meter Walk Test | 20 seconds
  The 10-Meter Walk Test is a commonly used measure for assessing walking speed. For the 10 Meter Walk Test, two end lines and two buffer lines were taped on the ground. Each end line was 14 m from the other and the each buffer line was 2 m from the end line. The time to walk the middle 10 m was recorded using a stopwatch.
Timed 25-feet Walk Test | 1 minutes
  People with multiple sclerosis are instructed to walk 25 feet as fast, but safely, as possible. This test is timed from the moment the patient crossed the start line and stopped when people with multiple sclerosis is crossed the finish line.
Six Minute Walk Test | 6 minutes
  It is used to measure gait performance. Participants are instructed to walk as far as they could over 6 min. The total distance that a people can walk was measured in meters.
3-meter Backward Walk Test | 10 seconds
  The 3-m course was determined and marked with black tape on the tile or wood surface. The test was started by asking participants to stand straight facing backward and to position their heels at the baseline level of the black tape. The examiner instructed the participants to walk backward rapidly, but as safely as possible. This test was performed with 3 trials, and the average time was expressed in seconds.
Dynamic Gait Index | 5 minutes
  This test is designed to test eight facets of gait, including gait on even surface, gait with changing speed, gait with head turns in vertical and horizontal planes, stepping over or around obstacles, gait with pivot turns, and stair ascent and descent. It is scored a four-point ordinal scale, ranging from 0 to 3. The best possible score on the dynamic gait index is a 24.
Multiple Sclerosis Walking Scale-12 | 2 minutes
  The Multiple Sclerosis Walking Scale-12 is a 12-item patient-rated measure of the impact of multiple sclerosis on walking. Each item is rated on a scale ranging between 1 (Not at all) and 5 (Extremely). The total MSWS-12 score is computed by subtracting the minimum possible score of 12 points from the participant's score (i.e., sum of the 12 item scores), dividing by the maximal score of 60 points, and then multiplying the result by 100. This lead to a possible range of MSWS-12 scores between 0 and 80.
Timed Up and Go Test | 15 seconds
  TUG is used to assess functional mobility. Participants are given verbal instruction to stand up from an armchair, walk forward 3 m, turn round, walk back towards the armchair and sit down. The time taken to complete is recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Canan Yucesan, Prof. Dr., Principal Investigator — Ankara University
Locations (1):
- Ankara University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang J, Xu J, An R. Effectiveness of backward walking training on balance performance: A systematic review and meta-analysis. Gait Posture. 2019 Feb;68:466-475. doi: 10.1016/j.gaitpost.2019.01.002. Epub 2019 Jan 3. PMID 30616175
- [Background] Rose DK, DeMark L, Fox EJ, Clark DJ, Wludyka P. A Backward Walking Training Program to Improve Balance and Mobility in Acute Stroke: A Pilot Randomized Controlled Trial. J Neurol Phys Ther. 2018 Jan;42(1):12-21. doi: 10.1097/NPT.0000000000000210. PMID 29232308
- [Background] Choi JY, Son SM, Park SH. A Backward Walking Training Program to Improve Balance and Mobility in Children with Cerebral Palsy. Healthcare (Basel). 2021 Sep 9;9(9):1191. doi: 10.3390/healthcare9091191. PMID 34574964
- [Background] Moon Y, Bae Y. Backward walking observational training improves gait ability in patients with chronic stroke: randomised controlled pilot study. Int J Rehabil Res. 2019 Sep;42(3):217-222. doi: 10.1097/MRR.0000000000000352. PMID 30998551
- [Background] Wang J, Yuan W, An R. Effectiveness of backward walking training on spatial-temporal gait characteristics: A systematic review and meta-analysis. Hum Mov Sci. 2018 Aug;60:57-71. doi: 10.1016/j.humov.2018.05.007. Epub 2018 May 24. PMID 29804040
- [Background] DeMark L, Fox EJ, Spigel PM, Osborne J, Rose DK. Clinical application of backward walking training to improve walking function, balance, and fall-risk in acute stroke: a case series. Top Stroke Rehabil. 2019 Oct;26(7):497-502. doi: 10.1080/10749357.2019.1641011. Epub 2019 Jul 16. PMID 31311448